CLINICAL TRIAL: NCT02463175
Title: A Randomized Controlled Pilot Study to Examine the Effects of Goal-directed Fluid Therapy on Post-operative Outcomes in Children Undergoing Scoliosis Repair
Brief Title: Effects of Goal-directed Fluid Therapy on Post-operative Outcomes in Children Undergoing Scoliosis Repair
Acronym: CardioQ-RP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with protocol compliance in both arms. Will simplify protocol.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Matthias Görges, PhD, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H14-03098
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Scoliosis; Acute Kidney Injury
Keywords: Fluid Therapy;; Transesophageal Doppler
MeSH Terms: conditions — Scoliosis; Acute Kidney Injury | interventions — Plasmalyte A; Crystalloid Solutions; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Fluid management, boluses of 5ml/kg of plasmalyte, will follow a specific goal-directed fluid therapy (GDT) protocol guided by transesophageal doppler measurement
  Interventions: Drug: Plasmalyte; Procedure: Goal-directed fluid therapy (GDT)
- Control group (Experimental): Fluid management, using boluses of 5ml/kg of plasmalyte, will follow the current standard of care guided by clinical judgment
  Interventions: Drug: Plasmalyte

INTERVENTIONS:
Drug: Plasmalyte — Boluses of 5ml/kg of plasmalyte
  Other Names: crystalloid solution for intravenous infusion
Procedure: Goal-directed fluid therapy (GDT) — Intraoperative goal-directed fluid therapy (GDT)
  Arms: Intervention group

SUMMARY:
Surgery for scoliosis correction, the abnormal curvature of the spine, is a major procedure often undertaken in adolescents. In adult anesthesia, there is a large volume of literature debating how to optimize fluids administered during surgery, as both too much fluid and too little fluid are associated with worse outcomes. The investigators will compare fluid administration based on the measured amount of blood pumped by the heart during each heart beat (goal-directed therapy), against standard anesthetic management. The main outcomes are a) post-surgical kidney dysfunction, b) prevalence of intraoperative hypotension, c) volumes of administered fluids, and d) length of hospitalization.

DETAILED DESCRIPTION:
1. Written informed consent from parent/guardian and assent from the patient will be obtained.
2. Each patient will be randomized into either the control arm or Cardio Q directed fluid therapy arm.
3. The following standard monitors will be placed before induction of anesthesia: electrocardiography, non-invasive blood pressure and pulse oximetry. The patient is anesthetized in the supine position using a standardized anesthetic technique. All attempts will be made to maintain normothermia
4. Following induction of anesthesia, the following will be placed: invasive arterial cannula, large bore intravenous cannula, Bispectral index monitor, temperature probe and central venous cannula (if needed).
5. Cardiac output monitor: Following induction of anesthesia and after placement of appropriate lines and monitors, a transoesophageal doppler (TED) probe will be inserted through the mouth into the esophagus and positioned correctly. A normal saline infusion will be started once the patient is anesthetized at 0.5 ml/kg/hour in the line where the drugs will be infused.

   1. Control Group: In this group, fluid administration, using boluses of 5ml/kg of plasmalyte at the anesthesiologist's discretion will be used. Anesthesiologists will be blinded to the cardio-Q numerics on the monitor. The flow waveform and sound will be available to optimize probe position.
   2. Intervention groups: Boluses of 5ml/kg plasmalyte will be given when: either MAP drops 20% from baseline or stroke volume drops 15% from baseline. If the patient is fluid responsive, a further 5ml/kg of fluid will be given.
   3. Vasopressor use: MAP (and stroke volume) becomes unresponsive to a fluid bolus then a bolus of phenylephrine or ephedrine may be given at the anesthesiologist's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scoliosis repair
* ASA physical status classification system (ASA) I-III

Exclusion Criteria:

* Pre-existing chronic kidney disease
* Oropharyngeal disease, e.g. pharyngitis
* Esophageal disease, e.g. heartburn, esophageal varices or hiatus hernia.
* Coagulopathy
* Scheduled for two stage procedures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postsurgical kidney dysfunction | Postop days 1-3
  Serum creatinine; urine output; urine based interleukin 18 (IL-18) and neutrophil gelatinase-associated lipocalin (NGAL) biomarkers

SECONDARY OUTCOMES:
Length of hospitalization | 30 days
Number of intra-operative hypotensive episodes | During surgery
  Number of MAP decrease below 75% of baseline reading in pre-anesthesia clinic
Percent case with intra-operative hypotension | During surgery
  Time spent hypotensive (MAP decrease below 75% of baseline reading) normalized by MAP measurement duration
Incidence of intra-operative spinal cord monitoring changes | During surgery
  From the neurological monitoring [when available]: motor evoked potentials (MEP) and somatosensory evoked potentials (SSEP)

CONTACTS AND LOCATIONS:
Overall Officials: Zoe E Brown, MBChB, FRCA, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada